CLINICAL TRIAL: NCT06105593
Title: Combined Effect of Balneotherapy and Physiotherapy Treatment in Female Infertility at Harkany Thermal Rehabilitation Centre: a Retrospective Study
Brief Title: Effect of Balneotherapy and Physiotherapy Treatment in Female Infertility: a Retrospective Study
Status: Active, not recruiting | Type: Observational
Sponsor: Harkány Thermal Rehabilitation Centre (Other)
Responsible Party: Sponsor
Other Study IDs: 9665-PTE 2023.
Record Dates: First submitted 2023-10-17; First posted 2023-10-27 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Infertility, Female
Keywords: Balneotherapy, Physiotherapy, Questionnaire, Infertility
MeSH Terms: conditions — Infertility, Female; Infertility

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to assess the effect of complex balneotherapy and physiotherapy treatment among infertile women treated in the Harkany Thermal Rehabilitation Center between July 01, 2007 and December 31, 2021. The main questions it aims to answer are:

* To what extent can the complex balneotherapy and physiotherapy treatment be an effective additional therapy in female infertility?
* What are the clinical changes behind infertility that can be helped by the complex balneotherapy and physiotherapy treatment? Participants will be asked to answer a questionnaire that we have prepared.

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* Diagnosed primary or secondary infertility

Exclusion Criteria:

* Lack of cooperation

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: In the period between July 1, 2007 and December 31, 2021, received a 3-week complex balneotherapy and physiotherapy treatment at the Harkany Thermal Rehabilitation Center in inpatient care
Sampling Method: Non-Probability Sample
Enrollment: 577 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
successful conception | 12 months
  Assessing with questionnaire. The participants are asked to answer the question whether they had a positive pregnancy test within 1 year after the complex balneotherapy and physiotherapy treatment at the Harkany Thermal Rehabilitation Center.

SECONDARY OUTCOMES:
successful delivery | 12 months
  Assessing with questionnaire. We ask the participants, if they managed to get pregnant within 1 year after the complex balneo and physiotherapy treatment to answer the question about what the outcome of their pregnancy was (for example: childbirth, miscarriage, stillbirth, etc.).
the effect of the treatments on successful conception in different causes of infertility | 12 months
  Assessing with questionnaire and statistical analysis. Based on the answers to the questionnaire, we will use statistical analysis to investigate the proportion of successful pregnancies after the complex balneotherapy and physiotherapy treatment in the case of the different pathologies underlying infertility.

CONTACTS AND LOCATIONS:
Overall Officials: Eszter Ambrus, Principal Investigator — Harkany Thermal Rehabilitation Center; Nóra Nusser, Study Director — Harkany Thermal Rehabilitacion Center
Locations (1):
- Harkany Thermal Rehabilitation Center, Harkány, Hungary

IPD SHARING:
Plan to Share IPD: No